CLINICAL TRIAL: NCT06947330
Title: Comparison Between Ultrasound Guided Erector Spinae Plane Block Versus Ultrasound Guided Serratus Anterior Plane Block Regarding Analgesia Post Modified Radical Mastectomy
Brief Title: Comparison Between Erector Spinae Plane Block Versus Serratus Anterior Plane Block Regarding Analgesia Post Modified Radical Mastectomy
Acronym: FMASUMD66/2025
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kholoud Usama (Other)
Responsible Party: Sponsor-Investigator, Kholoud Usama, Assistant Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FMASU-MD66/2025
Record Dates: First submitted 2025-04-13; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Modified Radical Mastectomy; Breast Cancer
Keywords: Breast Cancer; Modified Radical Mastectomy; Peripheral Nerve Block; Dexmedetomidine; Erector Spinae Plane Block; Serratus Anterior Plane Block; Ultrasound Guided; Adult Female
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Sampling method will be simple random. Patients will be randomly assigned into one of the following groups using opaque sealed envelopes:
  1. Group A (50 patients); will receive ultrasound guided Erector Spinae Plane Block.
  2. Group B (50 patients); will receive ultrasound guided Serratus Anterior Plane Block.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unilateral Erector Spinae group (Active Comparator): -The patient will be turned to the lateral decubitus position and the surgical side superiorly. After proper sterilization; The linear probe will be put in a parasagittal plane over the transverse process of thoracic 4 or thoracic 5 vertebrae, approximately 2.5 cm lateral to the spinous processes. The transverse process has a square form contour as compared to the rib which is rounded form contour. Then the 3 muscle layers or sheets with facial plane are distinguished from superficial to deep as trapezius, rhomboid major, and erector spinae with flickering pleura in between the transverse processes. The block will be managed unilaterally by in-plane technique using 22-gauge, 50 mm, echogenic needle which will be inserted in a cranial-caudal orientation and the block needle will be proceeded through the trapezius, rhomboid major, and erector spinae to smoothly contact the transverse process. Needle location will be confirmed by hydro-dissection on injecting 2-3 ml normal saline.
  Interventions: Procedure: Unilateral Erector Spinae group
- Unilateral Serratus Anterior group (Active Comparator): -After skin sterilization, with the patient in the lateral decubitus position and the side of surgery superiorly, the ultrasound linear probe will be put longitudinally oblique just below the mid-clavicle. After distinguish the second rib, the probe will be mobilized caudally and laterally (obliquely), towards the mid-axillary line to distinguish the third, fourth and fifth ribs. The ideal and definite probe position has its cephalad end at the anterior axillary line and the caudal end at the posterior axillary line. The facial plane between the serratus anterior muscle and ribs four and five will be identified between the 4th and 5th rib in the mid-axillary region. Under sonar guided, 50 mm echogenic needle will be advanced in-plane to introduce this facial plane in cranio-caudal direction.
  Interventions: Procedure: Unilateral Serratus Anterior group

INTERVENTIONS:
Procedure: Unilateral Erector Spinae group — On injecting 30 ml of bupivacaine 0.25% with 20 mcg Dexamedetomidine into the interfacial plane below erector spinae; a manifest linear pattern will be visualized uplifting the muscle.
  Other Names: Peripheral Nerve Block using Precedex; Erector Spinae block with Precedex as an adjuvant drug
  Arms: Unilateral Erector Spinae group
Procedure: Unilateral Serratus Anterior group — Once the needle will be in perfect position, confirmed by hydro-dissection on injecting 2-3 ml of normal saline, then 30 ml of bupivacaine 0.25% with 20 mcg Dexamedetomidine.
  Other Names: Peripheral Nerve Block using dexmedetomidine; Serratus Anterior Block with dexmedetomidine as an adjuvant drug
  Arms: Unilateral Serratus Anterior group

SUMMARY:
The goal of this clinical trial is to compare Ultrasound Guided Erector Spinae and Ultrasound Guided Serratus Anterior Plane Block post Modified Radical Mastectomy in adult females. the main questions it aims to answer are:

* Which of the two blocks has a better analgesic effect?
* Which of the two blocks is safer as regards inducing a pneumothorax and affecting the hemodynamics?

Participants:

* Will be divided into two groups after signing the informed consent.
* After being anesthetized and before surgical incision; the blocks will be given to the patient.
* Lung Ultrasound will be done for each patient to rule out pnemothorax once before the surgery and another after the end of surgery while the patient is being anesthetized.
* Patients that will experience pneuomothorax will be excluded from the study, and will be treated according to its size.
* Follow up of the patient for 24 hours postoperative to record the VAS score continuously, with giving increments of pethidine intravenously to relief pain.

DETAILED DESCRIPTION:
Breast surgeries belong to the most frequently performed procedures and are often associated with a high intensity of pain in the postoperative period.

Regional anesthesia techniques, have been the gold standard of postoperative pain management for breast surgeries. In recent years, the development of new techniques of regional anesthesia, which is due to the extensive implementation of ultrasound imaging, has enabled the use of a number of new blockades.The core mechanism of action in fascial blocks consists of blocking the nerve structures that supply a certain area of the trunk after deposition of local anesthetic within the fascial and fasciomuscular compartments. According to the current state of knowledge, the available options include Erector spinae plane block (ESPB) and Serratus anterior plane block (SAPB), however their recommendation in breast surgery requires more extensive scientific evidence.

Serratus anterior plane block acts on lateral branches of the intercostals nerves, blocking pain reception in the chest wall, while Erector spinae plane block involves the deposition of local anesthetic in the interfascial plane between erector spinae muscle and tips of the transverse processes of the vertebrae.

There is a scarcity of literature comparing ESPB and SAPB in patients undergoing breast surgeries.

Proponents of these techniques champion their ability to provide efficacious analgesia and anesthesia whereas critics cite a reportedly high failure rate and complications such as pneumothorax.

The German S3-guidelines suggest Lung Ultrasound as a possible alternative to Chest X-ray for the diagnosis of post-interventional pneumothorax.

Dexamedetomidine is a highly selective drug α2-adrenergic receptor agonist. Dexmedetomidine has the characteristics of sedation, analgesia, anti-anxiety, inhibition of sympathetic activity, mild respiratory inhibition, and stable hemodynamics. Numerous studies has revealed that dexmedetomidine in peripheral nerve blocks can shorten the onset time of anesthesia and prolong the time of sensory and motor nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status II, or III.
* Age 21 - 65 years.
* Female gender

Exclusion Criteria:

* ASA IV, V, VI.
* Infection at site of block.
* Coagulopathy, or patients on antiplatelets, or anticoagulants.
* Previous anesthetic allergy to bupivacaine.
* Distant organ metastasis.
* Male gender.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score for pain | at 0, 2, 4, 6, 8, 16, 20, 24 hours postoperatively
  * After extubation, the patient will be discharged from the operating room. VAS will be used to assess the postoperative pain (Myles et al., 2017).
  * Visual analogue scale score:
  Grade 0 (0-1 units on a scale): Good analgesia. Grade I (2-4 units on a scale): Moderate analgesia Grade II (5-7 units on a scale): Mild analgesia Grade III (8-10 units on a scale): No analgesia.
  * If VAS >3 units on a scale postoperatively, IV increment of pethidine 30 mg diluted in 5 ml saline will be given.
  * VAS ranging from (0 units on a scale) no pain, to (10 units on a scale) severe intolerable pain;

SECONDARY OUTCOMES:
Total dose of pethidine in mg. | at 0, 2, 4, 6, 8, 16, 20, 24 hours postoperatively
  If VAS >3 units on a scale postoperatively, IV increment of pethidine 30 mg diluted in 5 ml saline will be given.
Duration of analgesia postoperatively in hours. | at 0, 2, 4, 6, 8, 16, 20, 24 hours postoperatively
  If VAS >3 units on a scale postoperatively, IV increment of pethidine 30 mg diluted in 5 ml saline will be given.
Rate of vital data changes over the postoperative period | every 2 hour during the first 6 hours and then every 6 hours for 24 hours postoperatively.
  HR and MBP will be measured upon arrival to the PACU and after 30 min, then every hour if the patients remain in the PACU.
  In the surgical ward, vital signs (HR, SBP, MBP, DBP) as well as pain intensity will be assessed every 2 hour during the first 6 hours and then every 6 hours for 24 hours postoperatively.
Incidence of pneumothorax | Intra-operatively
  * Measurement tool: Lung ultrasound
  * After giving the block in each group, Lung Ultrasound will be performed on patients in the supine body position. The transducer will be placed longitudinally at the highest point of the anterior thorax, then moved along the intercotal spaces of the parasternal line and laterally, between the anterior and posterior axillary line, checking for lung sliding and lung point in 2D B-mode, and for seashore or stratosphere sign in M-mode. The hemithorax without intervention was examined first and then compared to the hemithorax with intervention.
  * The Lung Ultrasound will be repeated after the end of the surgery, while the patient is anesthetized, and before extubation. Cases of pneumothoraces either large or small will be excluded from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain-Shams University, Cairo, Waili, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Liu Z, Feng C, Jin Y, Zhao X. Dexmedetomidine as an Adjuvant in Peripheral Nerve Block. Drug Des Devel Ther. 2023 May 17;17:1463-1484. doi: 10.2147/DDDT.S405294. eCollection 2023. PMID 37220544
- [Background] Abd Elmohsen Bedewy A, Mohamed MS, Sultan HM, Khalil MS. Comparison Between Erector Spinae Plane Block versus Serratus Anterior Plane Block Regarding Analgesia and Stress Response After Modified Radical Mastectomy: Randomized Controlled Trial. Anesth Pain Med. 2024 Mar 26;14(2):e142189. doi: 10.5812/aapm-142189. eCollection 2024 Apr. PMID 38741901
- See also: Kumar, M.N., Begum, B.S. and R. Iniya (2022). A prospective randomized comparative study on erector spinae plane block and serratus anterior plane block in the postoperative pain management after breast surgeries. International Journal of Health Sciences — https://sciencescholar.us/journal/index.php/ijhs/article/view/10550
- See also: Gola, W., Białka, S., Andrzejewska, A., Palaczynski, P. and Misiołek, H. (2022). Fascial plane blocks for breast surgery - current state of knowledge. Anaesthesiology Intensive Therapy, [online] 54(3), pp.262-270. — https://pubmed.ncbi.nlm.nih.gov/36062421/
- See also: Mangold, M.S., Rüber, F., Steinack, C., Gautschi, F., Wani, J., Grimaldi, S. and Franzen, D.P. (2023). Lung Ultrasound for the Exclusion of Pneumothorax after Interventional Bronchoscopies-A Retrospective Study. Journal of Clinical Medicine, [online] 12( — https://pubmed.ncbi.nlm.nih.gov/36836009/
- See also: Muhammad, Q.U.A., Sohail, M.A., Azam, N.M., Bashir, H.H., Islam, H., Ijaz, R., Aquil, S., Mansoor, T., Dhakal, B., Fatima, T., Noor, J., Khan, A.S., Iqbal, A., Khatri, M. and Kumar, S. (2024). Analgesic efficacy and safety of erector spinae versus serrat — https://janesthanalgcritcare.biomedcentral.com/articles/10.1186/s44158-023-00138-y
- See also: Nair, A., &Diwan, S. (2022). Efficacy of ultrasound-guided serratus anterior plane block for managing pain due to multiple rib fractures: a scoping review. Cureus, 14(1). — https://pubmed.ncbi.nlm.nih.gov/35186581/
- See also: Ülgey, A., Pehlivan, S. S., &Demir, Ö. F. (2021). Postoperative thoracic pain treatment: serratus anterior or erector spinae plane block?. The Thoracic and Cardiovascular Surgeon, 69(06), 570-576. — https://pubmed.ncbi.nlm.nih.gov/33099765/
- Available data/document: Study Protocol — https://www.ilovepdf.com/download/6bhl069fp1wzcttl2h9kympvwcw0z348Az4p933p7tx6gm77hss9dbx3gbxjvm9ypjzwt97hdptj659jxht28ybgh1m4lyj34sth4k980tx1wzvm0A2pjghl7rs70r7pk67kblvbcfl9fn68lp5c06pjtdd07x9jqh7grqdl8b1kkp3b6271/88w